CLINICAL TRIAL: NCT06055478
Title: Effect of Ultrasound-guided Suprascapular Nerve Block and Axillary Nerve Block in Relieving Postoperative Pain After Arthroscopic Rotator Cuff Repair
Brief Title: Effect of Suprascapular Nerve Block and Axillary Nerve Block After Arthroscopic Rotator Cuff Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Collaborators: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2023-07-017-001
Record Dates: First submitted 2023-09-15; First posted 2023-09-26 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Rotator Cuff Tears
Keywords: suprascapular nerve block(SSNB); axillary nerve block(ANB); visual analog pain scale(VAS); patient's satisfaction(SAT); pain related cytokines; arthroscopic rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: Study group: Preemptive US guided suprascapular nerve block (SSNB) and axillary nerve block (ANB) using each 0.75% ropivacaine 10mL Control group: Preemptive US guided suprascapular nerve block (SSNB) and axillary nerve block (ANB) using each 0.9% saline 10mL
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent nurse uses a random number generator and allocates paticipants into the two group. Participant, investigator, and outcome assessor are blinded of the allocation information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preemptive ultrasound-guided suprascapular nerve block and axillary nerve block using ropivacaine (Experimental): Preemptive ultrasound-guided suprascapular nerve block and axillary nerve block using each 0.75% ropivacaine 10mL when arthroscopic rotator cuff repair Patient Controlled Analgesia (PCA) at a low fixed dose: fentanyl-loading dose: 0.4㎍/kg, continuous dose: 0.2㎍/kg/h, nefopam-loading dose: 0.04mg/kg, continuous dose: 0.02mg/kg/h
  Interventions: Procedure: Preemptive ultrasound-guided suprascapular nerve block and axillary nerve block
- Preemptive ultrasound-guided suprascapular nerve block and axillary nerve block using saline (Placebo Comparator): Preemptive ultrasound-guided suprascapular nerve block and axillary nerve block using each 0.9% saline 10mL when arthroscopic rotator cuff repair Patient Controlled Analgesia (PCA) at a low fixed dose: fentanyl-loading dose: 0.4㎍/kg, continuous dose: 0.2㎍/kg/h, nefopam-loading dose: 0.04mg/kg, continuous dose: 0.02mg/kg/h
  Interventions: Procedure: Preemptive ultrasound-guided suprascapular nerve block and axillary nerve block

INTERVENTIONS:
Procedure: Preemptive ultrasound-guided suprascapular nerve block and axillary nerve block — Preemptive ultrasound-guided suprascapular nerve block and axillary nerve block using ropivacaine or saline.
  Low fixed dose patient controlled analgesia (PCA) were done in the two group.
  Other Names: a low fixed dose patient controlled analgesia (PCA)

SUMMARY:
The goal of this clinical trial is to verify the effect of suprascapular nerve block and axillary nerve block in relieving postoperative pain after arthroscopic rotator cuff repair.

Are there differences in visual analog pain scale and patient's satisfaction? Are there differences in mean plasma pain related cytokines? The participants will undergo preemptive ultrasound guided suprascapular nerve block and axillary nerve block using each 0.75% ropivacaine 10mL or each 0.9% saline 10mL.

ELIGIBILITY:
Inclusion Criteria:

* a definite rotator cuff tear that needed repair seen on preoperative magnetic resonancce imaging (MRI)
* acceptance of arthroscopic surgery including rotator cuff repair
* age same as or more than 20 years
* acceptance of preemptive regional block and PCA, and blood testing

Exclusion Criteria:

* did not undergo arthroscopic rotator cuff repair
* stopped PCA before 48 hours postoperatively because of associated side effects
* a history of previous ipsilateral shoulder operation or fracture
* a concomitant neurologic disorder around the shoulder
* a failure of blood sampling including hemolysis, etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-09-18 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
visual analog pain scale (VAS) | preoperative, postoperative 1, 3, 6, 12, 18, 24, 36, 48 hour(s)
  0-10, 0: no pain, 10: very severe pain

SECONDARY OUTCOMES:
Patient's satisfaction (SAT) | preoperative, postoperative 1, 3, 6, 12, 18, 24, 36, 48 hour(s)
  0-10, 0: not satisfied, 10: very much satisfied
plasma Cortisol | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  ng/mL
IL-6 | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  pg/mL
IL-8 | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  pg/mL
IL-1β | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  pg/mL
Substance P | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  pg/mL
Serotonin | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  ng/mL
β -endorphin | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  pg/mL
norepinephrine | preoperative, postoperative 1, 6, 12, 24, 48 hour(s)
  pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Taek Hwang, MD,PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Jung-Taek Hwang, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No
We can decide it after the termination of this study.

REFERENCES:
- [Result] Lee JJ, Kim DY, Hwang JT, Song DK, Lee HN, Jang JS, Lee SS, Hwang SM, Moon SH, Shim JH. Dexmedetomidine combined with suprascapular nerve block and axillary nerve block has a synergistic effect on relieving postoperative pain after arthroscopic rotator cuff repair. Knee Surg Sports Traumatol Arthrosc. 2021 Dec;29(12):4022-4031. doi: 10.1007/s00167-020-06288-8. Epub 2020 Sep 25. PMID 32975624
- [Result] Lee JJ, Kim DY, Hwang JT, Lee SS, Hwang SM, Kim GH, Jo YG. Effect of ultrasonographically guided axillary nerve block combined with suprascapular nerve block in arthroscopic rotator cuff repair: a randomized controlled trial. Arthroscopy. 2014 Aug;30(8):906-14. doi: 10.1016/j.arthro.2014.03.014. Epub 2014 May 29. PMID 24880194